CLINICAL TRIAL: NCT06454318
Title: Screening Moderate to Severe Obstructive Sleep Apnea With Wearable Device
Status: Completed | Type: Observational
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, James Tisyakorn, Doctor, Thammasat University Hospital
Other Study IDs: MTU-EC-IM-1-066/65
Record Dates: First submitted 2024-04-13; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea; Polysomnography; Pulse Oximetry
Keywords: Obstructive Sleep Apnea; polysomnography; Pulse oximetry; ring-type pulse oximeter; wearable healthcare device
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Patients undergoing polysomnography and having Wellue O2 ring wear when doing polysomnography
  Interventions: Diagnostic Test: Wellue O2 ring

INTERVENTIONS:
Diagnostic Test: Wellue O2 ring — Wellue O2 ring wore when doing the polysomnography

SUMMARY:
The goal of this study is to find the best method to use Wellue O2 ring to screen for moderate to severe obstructive sleep apnea. The method that investigators use to screen for moderate to severe obstructive sleep apnea is oxygen desaturation index(ODI). The main questions of this study are

1. What is the best ODI to screen for moderate to severe obstructive sleep apnea?
2. What are the sensitivity, specificity and AUC of the study? In this study, participants are recruited from Sleep center of Thammasat prior to polysomnography. All participants in this study will

1. Undergo polysomnography according to Sleep center of Thammasat protocol 2. Wear Wellue O2 ring when undertaking polysomnography If the polysomnography is switch to PAP titration Wellue O2 ring will be taken out.

Data of Oxygen data from Wellue O2 ring are collected and compared with AHI. Investigators will find the best ODI to screen for obstructive sleep apnea.

DETAILED DESCRIPTION:
Background:

* Obstructive sleep apnea is a highly prevalent sleep-related disease.
* Moderate to severe obstructive sleep apnea is linked with traffic accident and other medical condition such as hypertension, pulmonary hypertension, myocardial infarction, stroke and diabetes mellitus
* Screening for obstructive sleep apnea using questionaires such as STOP-BANG and ESS (Epworth sleepiness scale) provide good sensitivity but low specificity
* Polysomnography used to diagnosed obstructive sleep apnea has limited assessibility and prolonged waiting time.
* Overnight pulse oximetry had been used to screen for obstructive sleep apnea and provided good sensitivity and specificity for screening obstructive sleep apnea using ODI (Oxygen desaturation index)
* Wellue O2 ring, a commercial grade pulse oximeter, with a frequency of measuring oxygen saturation of 0.25 Hz (compare to overnight pulse oximetry of 1 Hz) can measured oxygen saturation overnight with lower cost than overnight pulse oximetry (medical grade device)
* In this study, investigators want to find the best ODI to use to screen for moderate to severe obstructive sleep apnea. Investigators will find the sensitivity specificity and AUC of ROC curver in each ODI.

Outcome

* Sensitivity, Specificiy and area under the curve of ROC curve of each ODI. Sample size calculation
* Referencing previous studies (Kapur VK, Auckley DH, Chowdhuri S, et al. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017;13(3):479-504. Published 2017 Mar 15. doi:10.5664/jcsm.6506) The sensitivity of single channel home sleep test is 73% using Z = 1.96 and prevalence of 0.64 and d = 0.1 investigators get a population of 118 people. Investigators collected 42 more people in case of total sleep time < 2 hours.

Recruitment

* Patients are recruited prior to undertaking polysomnography test Eligibility criteria Inclusion criteria
* Patients age ≥ 18 years old Exclusion criteria
* Patients with pacemaker or intra-cardiac defibrillator
* Patients with suspected periodic limb movement disorder, insomnia, parasomnia, nacrolepsy and obesity hypoventilation syndrome
* Patients who canot wear O2 ring
* Patients with congestive heart failure, COPD, Asthma or Neuromuscular disorder
* Patients with desaturation when awake
* Patient with Scleroderma and Raynaud phenomenon

Study procedures

* After inform consent was obtained age, gender, body weight, height, neck circumference,underlying disease, STOP-BANG and ESS score are recorded
* Patients wear Wellue O2 ring when undergoing polysomnography, oxygen data were recorded from wellue O2 ring
* Data of AHI is extracted from the polysomnography report
* Data from wellue O2 ring is exported from wellu2 O2 ring using bluetooth in .csv format.
* Investigators excluded patient with Total sleep time < 2 hrs
* Baseline characteristic, oxygen saturation data and AHI are inputed in STATA version 17
* Investigators find the multiple ODI criteria and find the best ODI with the best sensitivity and specificity and AUC of ROC for screening moderate to severe obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Undertaking polysomnography at Sleep center of Thammasat

Exclusion Criteria:

* Patient with pacemaker or intra-cardiac defibrillator
* Patient suspected to have periodic limb movement disorder, insomnia, parasomnia, narcolepsy, obesity hypoventilation syndrome
* Patient who cannot wear Wellue O2 ring
* Patient suspected to have congestive heart failure, COPD, neuromuscular disorder
* Patient who have baseline O2 saturation below 92%
* Patient who have scleroderma or having Raynaud phenomenon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients whom undertaking polysomnography at Sleep center of Thammasat
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity | through study completion, an average of 1 year
  Sensitivity of each ODI
Specificity | through study completion, an average of 1 year
  Specificy of each ODI
AUC of ROC | through study completion, an average of 1 year
  Area under the curve of receiver operator curve of each ODI

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep center of Thammasat, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Neruntarat C, Chantapant S. Prevalence of sleep apnea in HRH Princess Maha Chakri Srinthorn Medical Center, Thailand. Sleep Breath. 2011 Dec;15(4):641-8. doi: 10.1007/s11325-010-0412-x. Epub 2010 Sep 17. PMID 20848319
- [Background] Stewart SA, Penz E, Fenton M, Skomro R. Investigating Cost Implications of Incorporating Level III At-Home Testing into a Polysomnography Based Sleep Medicine Program Using Administrative Data. Can Respir J. 2017;2017:8939461. doi: 10.1155/2017/8939461. Epub 2017 Jul 16. PMID 28790878
- [Background] Arias MA, Garcia-Rio F, Alonso-Fernandez A, Martinez I, Villamor J. Pulmonary hypertension in obstructive sleep apnoea: effects of continuous positive airway pressure: a randomized, controlled cross-over study. Eur Heart J. 2006 May;27(9):1106-13. doi: 10.1093/eurheartj/ehi807. Epub 2006 Feb 23. PMID 16497687
- [Background] Campos-Rodriguez F, Martinez-Garcia MA, Reyes-Nunez N, Caballero-Martinez I, Catalan-Serra P, Almeida-Gonzalez CV. Role of sleep apnea and continuous positive airway pressure therapy in the incidence of stroke or coronary heart disease in women. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1544-50. doi: 10.1164/rccm.201311-2012OC. PMID 24673616
- [Background] Fu Y, Xia Y, Yi H, Xu H, Guan J, Yin S. Meta-analysis of all-cause and cardiovascular mortality in obstructive sleep apnea with or without continuous positive airway pressure treatment. Sleep Breath. 2017 Mar;21(1):181-189. doi: 10.1007/s11325-016-1393-1. Epub 2016 Aug 8. PMID 27502205
- [Background] Gami AS, Pressman G, Caples SM, Kanagala R, Gard JJ, Davison DE, Malouf JF, Ammash NM, Friedman PA, Somers VK. Association of atrial fibrillation and obstructive sleep apnea. Circulation. 2004 Jul 27;110(4):364-7. doi: 10.1161/01.CIR.0000136587.68725.8E. Epub 2004 Jul 12. PMID 15249509
- [Background] George CF. Sleep apnea, alertness, and motor vehicle crashes. Am J Respir Crit Care Med. 2007 Nov 15;176(10):954-6. doi: 10.1164/rccm.200605-629PP. Epub 2007 Sep 6. PMID 17823357
- [Background] Gottlieb DJ, Yenokyan G, Newman AB, O'Connor GT, Punjabi NM, Quan SF, Redline S, Resnick HE, Tong EK, Diener-West M, Shahar E. Prospective study of obstructive sleep apnea and incident coronary heart disease and heart failure: the sleep heart health study. Circulation. 2010 Jul 27;122(4):352-60. doi: 10.1161/CIRCULATIONAHA.109.901801. Epub 2010 Jul 12. PMID 20625114
- [Background] Hla KM, Young T, Hagen EW, Stein JH, Finn LA, Nieto FJ, Peppard PE. Coronary heart disease incidence in sleep disordered breathing: the Wisconsin Sleep Cohort Study. Sleep. 2015 May 1;38(5):677-84. doi: 10.5665/sleep.4654. PMID 25515104
- [Background] Ismail K, Roberts K, Manning P, Manley C, Hill NS. OSA and pulmonary hypertension: time for a new look. Chest. 2015 Mar;147(3):847-861. doi: 10.1378/chest.14-0614. PMID 25732450
- [Background] Lavie P, Herer P, Hoffstein V. Obstructive sleep apnoea syndrome as a risk factor for hypertension: population study. BMJ. 2000 Feb 19;320(7233):479-82. doi: 10.1136/bmj.320.7233.479. PMID 10678860
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Martinez-Garcia MA, Campos-Rodriguez F, Catalan-Serra P, Soler-Cataluna JJ, Almeida-Gonzalez C, De la Cruz Moron I, Duran-Cantolla J, Montserrat JM. Cardiovascular mortality in obstructive sleep apnea in the elderly: role of long-term continuous positive airway pressure treatment: a prospective observational study. Am J Respir Crit Care Med. 2012 Nov 1;186(9):909-16. doi: 10.1164/rccm.201203-0448OC. Epub 2012 Sep 13. PMID 22983957
- [Background] Mehra R, Benjamin EJ, Shahar E, Gottlieb DJ, Nawabit R, Kirchner HL, Sahadevan J, Redline S; Sleep Heart Health Study. Association of nocturnal arrhythmias with sleep-disordered breathing: The Sleep Heart Health Study. Am J Respir Crit Care Med. 2006 Apr 15;173(8):910-6. doi: 10.1164/rccm.200509-1442OC. Epub 2006 Jan 19. PMID 16424443
- [Background] Tregear S, Reston J, Schoelles K, Phillips B. Obstructive sleep apnea and risk of motor vehicle crash: systematic review and meta-analysis. J Clin Sleep Med. 2009 Dec 15;5(6):573-81. PMID 20465027
- [Background] Yamakawa H, Shiomi T, Sasanabe R, Hasegawa R, Ootake K, Banno K, Wakayama H, Katada M, Kobayashi T. Pulmonary hypertension in patients with severe obstructive sleep apnea. Psychiatry Clin Neurosci. 2002 Jun;56(3):311-2. doi: 10.1046/j.1440-1819.2002.00957.x. PMID 12047610
- [Result] Chiu HY, Chen PY, Chuang LP, Chen NH, Tu YK, Hsieh YJ, Wang YC, Guilleminault C. Diagnostic accuracy of the Berlin questionnaire, STOP-BANG, STOP, and Epworth sleepiness scale in detecting obstructive sleep apnea: A bivariate meta-analysis. Sleep Med Rev. 2017 Dec;36:57-70. doi: 10.1016/j.smrv.2016.10.004. Epub 2016 Nov 5. PMID 27919588
- [Result] Nigro CA, Aimaretti S, Gonzalez S, Rhodius E. Validation of the WristOx 3100 oximeter for the diagnosis of sleep apnea/hypopnea syndrome. Sleep Breath. 2009 May;13(2):127-36. doi: 10.1007/s11325-008-0217-3. Epub 2008 Oct 2. PMID 18830731
- [Result] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- See also: Prevalence of sleep apnea in HRH Princess Maha Chakri Srinthorn Medical Center, Thailand — https://pubmed.ncbi.nlm.nih.gov/20848319/
- See also: Investigating Cost Implications of Incorporating Level III At-Home Testing into a Polysomnography Based Sleep Medicine Program Using Administrative Data — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5534303/
- See also: Pulmonary hypertension in obstructive sleep apnoea: effects of continuous positive airway pressure: a randomized, controlled cross-over study — https://pubmed.ncbi.nlm.nih.gov/16497687/
- See also: Role of sleep apnea and continuous positive airway pressure therapy in the incidence of stroke or coronary heart disease in women — https://pubmed.ncbi.nlm.nih.gov/24673616/
- See also: Meta-analysis of all-cause and cardiovascular mortality in obstructive sleep apnea with or without continuous positive airway pressure treatment — https://pubmed.ncbi.nlm.nih.gov/27502205/
- See also: Association of atrial fibrillation and obstructive sleep apnea — https://pubmed.ncbi.nlm.nih.gov/15249509/
- See also: Sleep apnea, alertness, and motor vehicle crashes — https://pubmed.ncbi.nlm.nih.gov/17823357/
- See also: Pulmonary hypertension in patients with severe obstructive sleep apnea — https://pubmed.ncbi.nlm.nih.gov/12047610/
- See also: Validation of the WristOx 3100 oximeter for the diagnosis of sleep apnea/hypopnea syndrome — https://pubmed.ncbi.nlm.nih.gov/18830731/
- See also: Diagnostic accuracy of the Berlin questionnaire, STOP-BANG, STOP, and Epworth sleepiness scale in detecting obstructive sleep apnea: A bivariate meta-analysis — https://pubmed.ncbi.nlm.nih.gov/27919588/
- See also: Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study — https://pubmed.ncbi.nlm.nih.gov/15781100/
- See also: Obstructive sleep apnoea syndrome as a risk factor for hypertension: population study — https://pubmed.ncbi.nlm.nih.gov/10678860/
- See also: Cardiovascular mortality in obstructive sleep apnea in the elderly: role of long-term continuous positive airway pressure treatment: a prospective observational study — https://pubmed.ncbi.nlm.nih.gov/22983957/
- See also: Coronary heart disease incidence in sleep disordered breathing: the Wisconsin Sleep Cohort Study — https://pubmed.ncbi.nlm.nih.gov/25515104/
- See also: OSA and pulmonary hypertension: time for a new look — https://pubmed.ncbi.nlm.nih.gov/25732450/
- See also: Association of nocturnal arrhythmias with sleep-disordered breathing: The Sleep Heart Health Study — https://pubmed.ncbi.nlm.nih.gov/16424443/
- See also: Prospective study of obstructive sleep apnea and incident coronary heart disease and heart failure: the sleep heart health study — https://pubmed.ncbi.nlm.nih.gov/20625114/
- See also: Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline — https://pubmed.ncbi.nlm.nih.gov/28162150/